CLINICAL TRIAL: NCT01017237
Title: Comparison of the Effectiveness of Sedation With i.v. Dexmedetomidine in Combination With Midazolam Alone or Midazolam and Low Dose Ketamine for Extraction of Third Molars.
Brief Title: Dexmedetomidine Sedation With Third Molar Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol proved to be ineffective for adequate sedation for third molar surgery.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-2157
Record Dates: First submitted 2009-08-14; First posted 2009-11-20 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2012-04

CONDITIONS: Anesthesia
Keywords: Dexmedetomidine sedation; Oral surgery sedation; Dexmedetomidine amnesia
MeSH Terms: interventions — Dexmedetomidine; Midazolam; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dex plus midazolam (Active Comparator): Dexmedetomidine loading dose of 0.4 mcg/kg followed by an infusion of 0.5 mcg/kg/hr plus midazolam 0.04 mg/kg i.v.
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam
- Dex plus midazolam and ketamine (Active Comparator): Dexmedetomidine loading dose of 0.4 mcg/kg followed by an infusion of 0.5 mcg/kg/hr plus midazolam 0.04 mg/kg and 0.25 mg/kg ketamine i.v.
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam; Drug: Ketamine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be infused at a rate of 6 mcg/kg/hr for four minutes; resulting in a loading dose of 0.4 mcg/kg, Followed by an infusion of 0.5 mcg/kg/hr will be initiated and continued until the completion of surgery.
  Other Names: Precedex
Drug: Midazolam — Midazolam 0.04 mg/kg i.v. administered after dexmedetomidine loading dose.
  Other Names: Versed
Drug: Ketamine — Ketamine 0.25 mg/ml administered i.v. following the dexmedetomidine loading dose and the midazolam.
  Other Names: Ketalar
  Arms: Dex plus midazolam and ketamine

SUMMARY:
Intravenous sedation is used frequently for the relief of pain and anxiety associated with oral surgical procedures performed under local anesthesia. The purpose of this study is to learn about patient and surgeon satisfaction with sedation using Dexmedetomidine in combination with midazolam alone or with midazolam plus low dose ketamine while having wisdom teeth removed.

The sedation produced by dexmedetomidine is unique in that it mimics natural sleep, a unique quality not shared by other drugs. Dexmedetomidine is often used in anesthesia in hospital operating rooms and has been approved by the US Food and Drug Administration for the use planned in this study.

DETAILED DESCRIPTION:
Subjects who have been screened medically and are scheduled for third molar surgery in the University of North Carolina (UNC)Oral and Maxillofacial Surgery (OMFS) clinic will be asked to volunteer for the study by the evaluating OMFS resident or attending physician. No additional x-rays will be taken other than those usually indicated for 3rd molar surgery. Informed consent will be obtained by study investigators.

Subjects will be instructed to fast for at least 8 hours prior to their appointment. Surgery will be performed in the Oral & Maxillofacial Surgery operating/sedation clinic where all monitoring equipment as well as emergency equipment is readily available, including the ability to ventilate the patient with oxygen (bag-mask), the ability to intubate, resuscitation drugs and equipment including a defibrillator. Patients will be positioned in a semi-reclining position in the dental chair and all monitors applied. A 20 gauge i.v. catheter will be placed and normal saline infusion attached. Supplemental oxygen will be administered via nasal cannula at 3 liters per minute. A picture will then be shown for recall testing. Pulse rate, arterial oxygen saturation (SpO2), respiratory rate, blood pressure, end-tidal CO2 (ETCO2), Ramsey Sedation Score (RSS sedation score) and Bispectral Index Scale (BIS) value will be recorded as a baseline and at 5 minute intervals during the procedure. Any SpO2 values below 90% as well as any episodes of apnea greater than 20 seconds will be recorded. Monitoring and recording of all data will be done by one of the investigators. Data will be recorded on pre-printed data forms. The surgical procedure will be performed by an oral and maxillofacial surgery resident physician.

Following the administration of 0.12 mg/kg of dexamethasone , dexmedetomidine will be infused at a rate of 6 mcg/kg/hr for four minutes; resulting in a loading dose of 0.4 mcg/kg. All of the above parameters will again be obtained and recorded. Patients will be randomly assigned by block randomization to receive either midazolam 0.04 mg/kg i.v. (50 patients), or midazolam 0.04 mg/kg plus 0.25 mg/kg of ketamine (50 patients). The operating surgeon and the patient will be blinded as to which protocol is being used. A dexmedetomidine infusion of 0.5 mcg/kg/hr will be initiated and continued until the completion of surgery. At this point local anesthesia will be administered in all four quadrants. Pain reaction during injections will be recorded. When efficacy of local anesthesia has been confirmed, surgery will commence. The surgery will be interrupted at 15 and 30 minutes to show a picture for recall testing by an investigator. If at any point the patient is deemed to be uncomfortable or uncooperative due to inadequate sedation, the protocol will be broken and additional sedation administered as per usual standards. The rescue therapy may include additional midazolam, ketamine, narcotic or propofol at the discretion of the anesthetist/sedationist. At the conclusion of surgery the dexmedetomidine infusion will be discontinued and the patient will be attended by a recovery nurse for collection of postoperative data. During recovery the physiologic parameters will be recorded at 10 minute intervals. When the patient achieves a recovery Aldrete score of >9, they will be asked by an investigator to recall pictures for amnesia assessment, and asked to assess patient satisfaction before leaving with an escort. The patient will be contacted on the day following surgery by phone or e-mail by one of the investigators to test for recall of pictures shown (amnesia testing) and patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status I and II
* Four asymptomatic third molars indicated for removal

Exclusion Criteria:

* Clinical history or ECG evidence of:

  * cardiac dysrhythmia or heart block
  * ischemic heart disease
  * asthma
  * sleep apnea
  * impaired liver, renal, or mental function
* chronic sedative or analgesic use
* allergies to any of the study drugs
* history of pericoronal infection with third molars

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay A Anderson, DDS, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina School of Dentistry, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients requiring extraction of third molars requiring sedation in the Oral Surgery clinic recruited.
Groups:
- Dex Plus Midazolam: Dexmedetomidine loading dose of 0.4 mcg/kg followed by an infusion of 0.5 mcg/kg/hr plus midazolam 0.04 mg/kg i.v.
  Dexmedetomidine : Dexmedetomidine will be infused at a rate of 6 mcg/kg/hr for four minutes; resulting in a loading dose of 0.4 mcg/kg, Followed by an infusion of 0.5 mcg/kg/hr will be initiated and continued until the completion of surgery.
  Midazolam : Midazolam 0.04 mg/kg i.v. administered after dexmedetomidine loading dose.
- Dex Plus Midazolam and Ketamine: Dexmedetomidine loading dose of 0.4 mcg/kg followed by an infusion of 0.5 mcg/kg/hr plus midazolam 0.04 mg/kg and 0.25 mg/kg ketamine i.v.
  Dexmedetomidine : Dexmedetomidine will be infused at a rate of 6 mcg/kg/hr for four minutes; resulting in a loading dose of 0.4 mcg/kg, Followed by an infusion of 0.5 mcg/kg/hr will be initiated and continued until the completion of surgery.
  Midazolam : Midazolam 0.04 mg/kg i.v. administered after dexmedetomidine loading dose.
  Ketamine : Ketamine 0.25 mg/ml administered i.v. following the dexmedetomidine loading dose and the midazolam.
Period: Overall Study
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Started | 10 | 8
Completed | 5 | 6
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Population: Total of 5 Dex plus midazolam subjects and 2 of 8 Dex plus midazolam plus ketamine sujects were disqualified and the protocol aborted due to lack of effect and uncooperative behavior requiring use of additional sedative agents
Groups:
- Total: Total of all reporting groups
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine | Total
Number analyzed (Participants) | 10 | 8 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 19 (3.6) | 20 (4.1) | 19 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Amnesia: Lack of Picture Recall Shown Prior to Sedation.
Description: Subjects were shown pictures of familiar objects prior to sedation, after the bolus dose of dexmedetomidine was administered, at 15 minutes and 30 minutes into the surgery and at the end of surgery. Subjects were shown a page containing multiple pictures to evaluate whether they could remember any of them. No recall demonstrating the presence of amnesia during that portion of the procedure. This process was repeated the day following surgery
Time Frame: Day of surgery prior to discharge
Population: Randomized per protocol
Measure: Number; unit: percentage of participants
Groups:
- Dexmedetomidine Plus Midazolam: Dexmedetomidine loading dose of 0.4 mcg/kg followed by an infusion of 0.5 mcg/kg/hr plus midazolam 0.04 mg/kg i.v.
  Dexmedetomidine : Dexmedetomidine will be infused at a rate of 6 mcg/kg/hr for four minutes; resulting in a loading dose of 0.4 mcg/kg, Followed by an infusion of 0.5 mcg/kg/hr will be initiated and continued until the completion of surgery.
  Midazolam : Midazolam 0.04 mg/kg i.v. administered after dexmedetomidine loading dose.
- Dexmedetomidine Plus Midazolam and Ketamine: Dexmedetomidine loading dose of 0.4 mcg/kg followed by an infusion of 0.5 mcg/kg/hr plus midazolam 0.04 mg/kg and 0.25 mg/kg ketamine i.v.
  Dexmedetomidine : Dexmedetomidine will be infused at a rate of 6 mcg/kg/hr for four minutes; resulting in a loading dose of 0.4 mcg/kg, Followed by an infusion of 0.5 mcg/kg/hr will be initiated and continued until the completion of surgery.
  Midazolam : Midazolam 0.04 mg/kg i.v. administered after dexmedetomidine loading dose.
  Ketamine : Ketamine 0.25 mg/ml administered i.v. following the dexmedetomidine loading dose and the midazolam.
Arm/Group | Dexmedetomidine Plus Midazolam | Dexmedetomidine Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
percentage of participants | 0 | 0

2. Secondary Outcome: Respiratory Parameters: Respiratory Rate
Description: Respirations per minute
Time Frame: Immediately prior to sedation
Population: Randomized per protocol
Measure: Mean (Standard Deviation); unit: Breaths per Minute
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
Breaths per Minute | 15 (3) | 17.2 (4)

3. Secondary Outcome: Respiratory Parameters: Respiratory Rate
Description: Rate of respirations
Time Frame: During surgical procedure
Population: per protocol
Measure: Mean (Standard Deviation); unit: Breaths per Minute
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
Breaths per Minute | 15 (3) | 19 (4)

4. Secondary Outcome: Respiratory Parameters: Oxyhemoglobin Saturation
Description: Oxyhemoglobin saturation per pule oximeter
Time Frame: Immediately prior to surgery
Population: per protocol
Measure: Mean (Standard Deviation); unit: Percent oxyhemoglobin saturation
Groups:
- Dex Plus Midazolam: Dexmedetomidine loading dose of 0.4 mcg/kg followed by an infusion of 0.5 mcg/kg/hr plus midazolam 0.04 mg/kg.
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
Percent oxyhemoglobin saturation | 98 (2.5) | 98 (2.4)

5. Secondary Outcome: Respiratory Parameters: Oxyhemoglobin Saturation
Description: Oxyhemoglobin saturation per pulse oximetry
Time Frame: During surgical procedure
Population: per protocol
Measure: Mean (Standard Deviation); unit: Percent oxyhemoglobin saturation
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
Percent oxyhemoglobin saturation | 98 (2.5) | 98 (3.4)

6. Primary Outcome: Amnesia: Lack of Recall One Day After Surgery of The Picture That Was Shown Prior to Sedation.
Description: Lack of recall of picture shown indicates presence of amnesia the day following surgery.
Time Frame: One day after surgery
Population: Per protocol
Measure: Number; unit: percentage of patients
Arm/Group | Dexmedetomidine Plus Midazolam | Dexmedetomidine Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
percentage of patients | 0 | 0

7. Primary Outcome: Amnesia: Lack of Picture Recall Following Dexmedetomidine Infusion Plus Midazolam.
Description: Percentage of patients unable to recall picture
Time Frame: Day of Surgery prior to discharge
Population: Per protocol
Measure: Number; unit: percentage of patients
Arm/Group | Dexmedetomidine Plus Midazolam | Dexmedetomidine Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
percentage of patients | 100 | 100

8. Primary Outcome: Amnesia: Lack of Recall One Day After Surgery of The Picture That Was Shown Following Dexmedetomidine Infusion Plus Midazolam.
Description: Inability to recall picture shown at this time indicates presence of amnesia on the day following surgery.
Time Frame: One day after surgery
Population: per protocol
Measure: Number; unit: percentage of patients
Arm/Group | Dexmedetomidine Plus Midazolam | Dexmedetomidine Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
percentage of patients | 100 | 100

9. Primary Outcome: Amnesia: Lack of Picture Recall Shown 15 Minutes Into Surgery
Description: Lack of recall of picture shown at this time indicates presence of amnesia
Time Frame: Day of Surgery prior to discharge
Population: per protocol
Measure: Number; unit: percentage of patients
Arm/Group | Dexmedetomidine Plus Midazolam | Dexmedetomidine Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
percentage of patients | 100 | 100

10. Primary Outcome: Amnesia: Lack of Recall One Day After Surgery of The Picture That Was Shown 15 Minutes Into Surgery.
Description: Lack of recall of picture demonstrates presence of amnesia on day following surgery
Time Frame: One day after surgery
Population: per protocol
Measure: Number; unit: percentage of patients
Arm/Group | Dexmedetomidine Plus Midazolam | Dexmedetomidine Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
percentage of patients | 100 | 100

11. Primary Outcome: Amnesia: Lack of Picture Recall Shown 30 Minutes Into Surgery
Description: Lack of recall of picture shown indicates presence of amnesia
Time Frame: Day of Surgery prior to discharge
Population: per protocol
Measure: Number; unit: percentage of patients
Arm/Group | Dexmedetomidine Plus Midazolam | Dexmedetomidine Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
percentage of patients | 83 | 100

12. Primary Outcome: Primary Title: Amnesia: Lack of Recall One Day After Surgery of The Picture That Was Shown 30 Minutes Into Surgery.
Description: Lack of recall of picture shown indicates presence of amnesia on day following surgery.
Time Frame: One day after surgery
Population: Per protocol
Measure: Number; unit: percentage of patients
Arm/Group | Dexmedetomidine Plus Midazolam | Dexmedetomidine Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
percentage of patients | 83 | 100

13. Primary Outcome: Amnesia: Lack of Picture Recall at Surgery End Time.
Description: Lack of recall of picture shown indicates presence of amnesia
Time Frame: Day of surgery prior to discharge
Population: per protocol
Measure: Number; unit: percentage of patients
Arm/Group | Dexmedetomidine Plus Midazolam | Dexmedetomidine Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
percentage of patients | 83 | 100

14. Primary Outcome: Amnesia: Lack of Recall One Day After Surgery of The Picture That Was Shown at Surgery End Time.
Description: Lack of recall of picture shown indicates presence of amnesia on day following surgery.
Time Frame: One day after surgery
Population: per protocol
Measure: Number; unit: percentage of patients
Arm/Group | Dexmedetomidine Plus Midazolam | Dexmedetomidine Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
percentage of patients | 83 | 100

15. Secondary Outcome: Respiratory Parameters: End-tidal Carbon Dioxide
Description: Measured via capnography at nares
Time Frame: Immediately prior to sedation
Population: per protocol
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
mmHg | 39.4 (4.7) | 36.2 (5.3)

16. Secondary Outcome: Respiratory Parameters: End-tidal Carbon Dioxide
Description: Measured by capnography at nares
Time Frame: Duration of surgery
Population: per protocol
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
mmHg | 36.9 (5.1) | 38.2 (4.76)

17. Secondary Outcome: Mean Arterial Blood Pressure
Description: Blood pressure per automated monitor
Time Frame: Immediately prior to surgery
Population: per protocol
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
mmHg | 96.2 (12.4) | 96.4 (15.3)

18. Secondary Outcome: Mean Arterial Blood Pressure
Description: Measured using automated blood pressure monitor
Time Frame: During duration of surgery
Population: per protocol
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
mmHg | 93.8 (21.2) | 95.9 (18.9)

19. Secondary Outcome: Heart Rate
Description: Heart rate per EKG monitor
Time Frame: Prior to sedation
Population: per protocol
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
Beats per minute | 66.8 (11.2) | 71.4 (18.4)

20. Secondary Outcome: Heart Rate
Description: Per EKG monitor
Time Frame: Duration of surgery
Population: per protocol
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
Beats per minute | 75 (12.4) | 85.6 (15.1)

21. Secondary Outcome: Surgeon Satisfaction With Sedation Technique
Description: Numerical value on scale of 1-5 from Very dissatisfied (1) to Extremely satisfied (5)
Time Frame: After surgery completed: day of surgery, within 15 minutes
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
units on a scale | 4.0 (0.4) | 3.2 (0.6)

22. Secondary Outcome: Patient Satisfaction With Sedation Technique
Description: Rating of how satisfied the patient was with their sedation on a scale of 1-5 with 1 being very dissatisfied and 5 being extremely satisfied
Time Frame: after completion of surgery (within 15 minutes)
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
units on a scale | 4.7 (0.2) | 4.8 (0.2)

23. Secondary Outcome: Ramsey Sedation Scale Score
Description: Rating of depth of sedation by sedationist. Scale 1 - 6, 1 being widw awake and 6 being non-responsive
Time Frame: During surgical procedure
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
units on a scale | 3.2 (0.4) | 3.5 (0.5)

24. Secondary Outcome: Bispectral Index Score (BIS)
Description: Bispectral Index (BIS) measures level of consciousness by algorithmic analysis of the patient's electroencephalogram (EEG) during anesthesia and sedation. The BIS can range from 0 (equivalent to EEG silence) to 100 (equivalent to fully awake and alert). A BIS value of 40-60 indicates an adequate general anesthesia state.
Time Frame: During surgery duration.
Population: per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Number analyzed (Participants) | 5 | 6
units on a scale | 75.1 (11.2) | 82.6 (12.4)

ADVERSE EVENTS:
Arm/Group | Dex Plus Midazolam | Dex Plus Midazolam and Ketamine
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

LIMITATIONS AND CAVEATS:
Early termination due to ineffective sedation. We had to abandon the protocol in 5 of 10 patients in the dexmedetomidine plus midazolam group and 2 of 8 patients in the dexmedetomidine plus midazolam and ketamine group because of combative behavior.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes